CLINICAL TRIAL: NCT05550012
Title: Evaluation of a New Deep-learning Based Artificial Intelligence Iterative Reconstruction (AIIR) Algorithm in Different Enhancement Phases of Low-dose Liver CT
Brief Title: A New Deep-learning Based Artificial Intelligence Iterative Reconstruction (AIIR) Algorithm in Low-dose Liver CT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Qingshi Zeng, Clinical Professor, Qianfoshan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: LD-SH-2022
Record Dates: First submitted 2022-09-14; First posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Deep Learning

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard-dose CT (No Intervention): those patients undergo standard-dose liver CT in portal vein and delayed phase
- low-dose CT (Experimental): those patients undergo low-dose liver CT in portal vein and delayed phase
  Interventions: Other: low-dose CT

INTERVENTIONS:
Other: low-dose CT — those patients undergo low-dose liver CT in portal vein and delayed phase.
  Arms: low-dose CT

SUMMARY:
CT-enhanced scans are routine imaging modality for the diagnosis and follow-up of liver disease. However, this means that patients will receive more radiation dose. Therefore, it is necessary to reduce the radiation dose received by patients as much as possible. Deep learning-based reconstruction algorithms have been introduced to improve image quality recently. For many years, researchers attempt to maintain image quality using an advanced method while reducing radiation dose. Recently, a new deep-learning based iterative reconstruction algorithm, namely artificial intelligence iterative reconstruction (AIIR, United Imaging Healthcare, Shanghai, China) has been introduced. In this study, we evaluate the image and diagnostic qualities of AIIR for low-dose portal vein and delayed phase liver CT with those of a KARL method normally used in standard-dose CT.

DETAILED DESCRIPTION:
In our hospital, patients with abdominal pelvic cancer undergo follow-up low-dose CT for the evaluation of treatment plan after clinical treatment or disease progress. The raw-data of low-dose CT were collected retrospectively and reconstructed using KARL and AIIR algorithm. In this study, we evaluate the image and diagnostic qualities of AIIR for low-dose portal vein and delayed phase liver CT with those of a KARL method normally used in standard-dose CT.

ELIGIBILITY:
Inclusion Criteria:

* those scheduled for contrast-enhanced liver CT

Exclusion Criteria:

* images affected by artifacts (motion or implants)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-09-30 (Estimated); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
signal-to-noise ratio (SNR) | 6 months
  Evaluate the image qualities of AIIR for low-dose portal vein and delayed phase liver CT with those of a KARL method normally used in standard-dose CT
contrast to noise ratio (CNR) | 6 months
  Evaluate the image qualities of AIIR for low-dose portal vein and delayed phase liver CT with those of a KARL method normally used in standard-dose CT
diagnostic confidence | 6 months
  Evaluate the diagnostic qualities of AIIR for low-dose portal vein and delayed phase liver CT with those of a KARL method normally used in standard-dose CT

CONTACTS AND LOCATIONS:
Overall Officials: Qingshi Zeng, Study Director — Qianfoshan Hospital
Locations (1):
- Qianfoshan Hospital (The First Affiliated Hospital of Shandong First Medical University), Jinan, Shandong, China